NCT number: [2021]075

## A multicenter randomized controlled trial of low-dose single-wavelength red light in the decrease of myopia incidence rate in the setting of school

Shanghai Eye Disease Prevention and Treatment Center

March 27, 2021

A multicenter randomized controlled trial of low-dose single-wavelength red light in the decrease of myopia incidence rate in the setting of school.

| Study aims and | l rationales | A multicenter randomized controlled trial exploring the effectiveness of low-dose single-wavelength red light on the prevention of myopia and the decrease of myopia incidence rate in children of grade 1-4 of primary schools (age of 6-12 years). |
|---|---|---|
| Primary aim | | To examine the effectiveness of low-dose single-wavelength red light on<br>the prevention of myopia and the decrease of myopia incidence rate in the<br>setting of school. |
| Secondary aim | | To examine the effect of low-dose single-wavelength red light on spherical equivalent (SE) and uncorrected visual acuity in school-aged children who are in pro-myopia status. |
| Study design | | A multicenter randomized controlled trail. |
| Study participa enrollment | nts and estimated | Primary school students of grade 1-4 who are in pro-myopia status will be enrolled as study participants. |
| 3. | | <ol> <li>Students of grade 1-4 in the participating schools;</li> <li>Students who are in pro-myopia status, as defined as cycloplegic SE between -0.5D(exclusive) and 0.5D (inclusive);</li> <li>Students whose mother and/or father are in myopia status (SE≤-3.0D for either of eyes);</li> <li>Students whose parents sign informed consent and agree to let their kids participate in study.</li> </ol> |
| Exclusion crite | | <ol> <li>Students whose parents do not sign informed consent;</li> <li>Students who have strabismus and/or other binocular vision abnormality;</li> <li>Students who have other eye diseases and/or systematic diseases</li> <li>Students who meet the standards with which investigators and study physicians think it is not appropriate to enroll.</li> </ol> |
| Sample size | | A total of 534 students will be included in the study, half of which(267) in the intervention group and half in the control group |
| Arrangement fo | | Baseline ophthalmic examinations will be conducted in March 2021; a total of three times of follow-ups will be administered in June, September and December 2021; end-point examinations will be conducted in march 2022. |
| Trial duration | | The trial will last 12 months starting from the baseline in March 2021 to the end point in March 2022. |
| Intervention | Intervention group | The enrolled students will be first stratified according to grade within each of the participating schools; within each of the stratified grade, the students will be randomly assigned in a ratio of 1:1 to either the intervention group or the control group. |
| | | Participants in the intervention group will receive low-dose single-wavelength red light intervention in the setting of school from the first day to the fifth day of the week; on summary and winter vocations, the participants will receive intervention at home every day. |

| | | The intervention lasts three minutes one time, two times a day, the interval between two exposures in a day should be more than 4 hours. |
|---|---|---|
| | Control group | Participants in the control group will not receive the intervention. |
| | | The cumulative incidence rate of myopia among intervention and control |
| Primary outcome | | groups. |
| Statistical hypothesis | | The intervention of low-dose single-wavelength red light can prevent myopia and decrease the incidence rate of myopia. |
| | | School-aged children, low-dose single-wavelength red light, prevention of |
| Key words | | myopia. |
| Supplementary information | | None. |